CLINICAL TRIAL: NCT01256905
Title: Attention Modulation for Treatment of Parkinson's Disease and Dementia With Lewy Bodies
Acronym: Armodafinil
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI departure from institution
Sponsor: NYU Langone Health (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0189
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Parkinsons Disease; Lewy Bodies Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Armodafinil (Experimental)
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — Armodafinil 150 mg

SUMMARY:
The purpose of this study is to evaluate if a drug commonly used to treat excessive day-time sleepiness, called armodafinil (Nuvigil), is also effective in improving the impairment in the attention commonly reported by patients with more advanced Parkinson's disease (PD) and Lewy body disease (LBD).

DETAILED DESCRIPTION:
The main aims of this study are:

1. To investigate whether in PDD and DLB th specific disturbances in the basal ganglia thalamocortical network, measured through the Electroencephalography (EEG) frequency analysis, are ameliorated by armodafinil.

Our main hypothesis is that armodafinil can restore the attention and improve cognitive disturbances in PDD and DLB, through a specific effect on striatal-thalamo-cortical activity.

ELIGIBILITY:
Inclusion Criteria:

* Established criteria for diagnosis of PDD (Parkinsons Disease) {Emre M et al. Mov Disord 2007;22:1689-707} and DLB (Lewy Bodies Disease) {McKeith et al. Neurology 2005;65:1863-72}
* Mini Mental State Examination (MMSE) score between <24; and/or Dementia Rating
* Scale-2 (DRS-2) score <134;
* Clinical Assessment of Fluctuation (CAF)>4;
* Stable anti-parkinsonian medication in the 4 weeks preceding the study

Exclusion Criteria:

* Use of cognitive enhancers (Donepezil, Rivastigmine, Galantamine, Modafinil, Memantine) in the last 4 weeks:

Concomitant use of any medication contraindicated with modafinil/armodafinil; History of alcohol and substances abuse. Use of medications known to alter the normal EEG activity in humans during the study period (i.e. clonazepam) History of psychiatric disorders, other than depression and psychiatric complication of PDD and DLB

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2011-08-08 (Actual); Study Completion 2011-08-08 (Actual)

PRIMARY OUTCOMES:
EGI netstation software (Electrical Geodesics Inc.) and a custom made software that runs on the Matlab platform (The Mathworks) | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sara Varanese, MD, Principal Investigator — NYU Parkinsons and Movement Disorders Center
Locations (1):
- NYU Parkinsons and Movement Disorders Center, New York, New York, United States

REFERENCES:
- See also: armodafinil — http://parkinson.med.nyu.edu/